CLINICAL TRIAL: NCT05629403
Title: Women's Hospital of Nanjing Medical University
Brief Title: Exclusive Breastfeeding Improves Puerperal Glucose Metabolism in Pregnant Women With Gestational Diabetes Mellitus and Links to Lipids Composition
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xirong Guo, Professor, Nanjing Medical University
Other Study IDs: NanjingMU2022
Record Dates: First submitted 2022-07-07; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Gestational Diabetes; Breast Feeding; Lipid Metabolism Disorders
MeSH Terms: conditions — Diabetes, Gestational; Breast Feeding; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exclusive breastfeeding: breastfeeding exclusively
  Interventions: Other: observe
- formula feeding: formula feeding
  Interventions: Other: observe

INTERVENTIONS:
Other: observe — no intervention

SUMMARY:
Breastfeeding could effectively be associated with a lower risk of future type 2 diabetes (T2D) in women with gestational diabetes mellitus (GDM), but the short-term protective impact of puerperal breastfeeding on maternal metabolic recovery of GDM women remains unascertained. The investigators recruited GDM participants at 6-9 weeks postpartum and retrieved clinical diagnoses of GDM from electronic medical records. Feeding patterns were collected via phone calls. Glucose metabolism parameters and lipid profiling were performed on fasting plasma samples collected from patients 6-9 weeks postpartum (20 breastfeeding cases vs. 15 formula feeding cases).

ELIGIBILITY:
Inclusion Criteria:

1. 18-35 years old;
2. gestational age greater than 37 weeks;
3. Body Mass Index (BMI) before pregnancy 18.5-28kg/m2;
4. Have normal listening and speaking skills, can communicate, and are willing to participate in this study.

Exclusion Criteria:

1. abnormal glucose metabolism or diabetes has been diagnosed before pregnancy;
2. assisted reproduction;
3. GDM patients requiring drug treatment;
4. The use of blood lipid regulation drugs;
5. other pregnancy complications and complications;
6. Suffering from heart, malignant tumor, kidney and other major organ diseases;
7. associated with neurological dysfunction and cognitive impairment;
8. Failure to cooperate with follow-up observers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women (aged 18-35 years) who delivered live-born infants equal to or greater than 37 weeks of gestation at the Women's Hospital of Nanjing Medical University (Nanjing, China) and were not using medications affecting glucose tolerance, lipid regulation and not planning another pregnancy within the next 2 years were enrolled. All the participants received 75g OGTT at 24-28 weeks of gestation and were diagnosed with GDM based on the IADPSG criteria (International Association of Diabetes and Pregnancy Study Groups Consensus Panel et al.). At 6-8 weeks postpartum, all the participants were administered regularly for a post-natal health check-up to classify the body and genitals basically restored status. Fasting plasma samples were collected to measure plasma glucose, and insulin, and reclassify glucose metabolic status. Frequency and amount of breastmilk feeding and formula feeding for each woman were evaluated by trained research staff via telephone calls.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
glucose | At 6-8 weeks postpartum
  glucose (mmol/L) determined with human ELISA kits
insulin | At 6-8 weeks postpartum
  insulin (mU/L) determined with human ELISA kits
c-peptide | At 6-8 weeks postpartum
  c-peptide (ng/m) determined with human ELISA kits
HOMA-IR | At 6-8 weeks postpartum
  fasting glucose and fasting glucose will be combined to report HOMA-IR

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Maternal and child Health Care Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No